CLINICAL TRIAL: NCT01700582
Title: French National Observatory of the Patients With Non-small Cell Lung (NSCLC) Benefiting From a Molecular Test on the Hospital Platforms of Molecular Genetics.
Brief Title: French National Observatory of the Patients With Non-small Cell Lung (NSCLC) and Molecular Testings
Status: Completed | Type: Observational
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Other Study IDs: Biomarkers-France
Record Dates: First submitted 2012-08-01; First posted 2012-10-04 (Estimated); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung; ALK Gene Mutation; KRAS Gene Mutation; BRAF Gene Mutation
Keywords: lung cancer; biomarkers; EGFR; KRAS; ALK; HER2; PI3K; BRAF; IFCT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with advanced lung cancer: Patients with advanced lung cancer

SUMMARY:
The French National Cancer Institute (INCa) support a 28 hospital platforms network for molecular testing of cancer patients. These platforms routinely assess a panel of biomarkers in order to speed up access of French cancer patients to targeted therapies (commercially available or through clinical trials).

The objective of the BIOMARKERS-France study is to describe the epidemiological, clinical and molecular characteristics of these patients and their tumors and to assess the impact of these analyzes on their treatment (ie bio-guided therapy) as well as outcomes (response rate, progression free and overall survival).

DETAILED DESCRIPTION:
The French National Cancer Institute (INCa) support a 28 hospital platforms network for molecular testing of cancer patients. These platforms routinely assess a panel of biomarkers in order to speed up access of French cancer patients to targeted therapies (commercially available or through clinical trials).

Regarding stage IV non-squamous NSCLC patients, 7 biomarkers are assessed including activating EGFR mutations, EML4-ALK translocation and EGFR T790M, KRAS, BRAF, HER2 and PI3KCA mutations. In 2012, up to 17 to 20,000 patients will be tested on this platform network.

The objective of the BIOMARKERS-France study is to describe the epidemiological, clinical and molecular characteristics of these patients and their tumors and to assess the impact of these analyzes on their treatment (ie bio-guided therapy) as well as outcomes (response rate, progression free and overall survival).

This study will collect, in a prospective way, data from a unique national cohort in order to guide future decisions regarding biomarker assessments (type? Number? Methods? Etc) in connexion with all the other research works currently ongoing in France.

ELIGIBILITY:
Inclusion Criteria:

* Advanced Non-small cell lung cancer (NSLC)
* Biomarkers analysis on hospital platforms

Exclusion Criteria:

- Histology other than NSLC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced non-small cell cancer
Sampling Method: Non-Probability Sample
Enrollment: 17664 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
EGF-R gene mutation in nationwide cohort | 1 Year
  Number of patients with EGF-R gene mutation

SECONDARY OUTCOMES:
K-RAS gene mutation in nationwide cohort | 1 year
  Number of patients with K-RAS gene mutation
EML4-ALK translocation in nationwide cohort | 1 year
  Number of patients with EML4-ALK translocation
BRAF gene mutation in nationwide cohort | 1 year
  Number of patients with BRAF gene mutation
HER2 gene mutation in nationwide cohort | 1 year
  Number of patients with HER2 gene mutation
PI3K gene mutation in nationwide cohort | 1 year
  Number of patients with PI3K gene mutation

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Barlesi, PhD, MD, Principal Investigator — IFCT, Aix Marseille Université / Assistance Publique Hôpitaux de Marseille
Locations (133):
- France (133):
  - Clinique Calabet - Centre de Radiothérapie et d'Oncologie, Agen
  - Clinique Claude Bernard, Albi
  - Clinique de l'Europe, Amiens
  - CHU d'Angers, Angers
  - Hôpital Privé d'Antony, Antony
  - CHIC, Aulnay-sous-Bois
  - Auxerre - CH, Auxerre
  - CH d'Avignon, Avignon
  - CH de la Côte Basque, Bayonne
  - CHU Besancon - Pneumologie, Besançon
  - CH de Béziers, Béziers
  - Blois - CH, Blois
  - CHU Avicenne, Bobigny
  - Hôpital Ambroise Paré - Pneumologie, Boulogne
  - Hôpital Fleyriat, Bourg-en-Bresse
  - Hôpital de Briançon, Briançon
  - CHU Côte de Nâcre, Caen
  - Cahors - CH, Cahors
  - CH de Cannes, Cannes
  - Chambray Les Tours - Clinique Léonard de Vinci, Chambray-lès-Tours
  - CH de Chartres Hôpital Louis Pasteur, Chartres
  - Chevilly-Larue - CH, Chevilly-Larue
  - Hôpital de Cholet - Pneumologie, Cholet
  - Hôpital Percy-Armées - Pneumologie, Clamart
  - Hôpital Pasteur, Colmar
  - Clinique des Cèdres, Cornebarrieu
  - Créteil - CHI, Créteil
  - Dax - CH, Dax
  - Denain - CH, Denain
  - Dijon - CAC, Dijon
  - Dijon - CHU, Dijon
  - Draguignan - CH, Draguignan
  - CH de Dreux, Dreux
  - Elbeuf - CH, Elbeuf
  - Ermont - Clinique Claude Bernard, Ermont
  - Epinal - CH, Épinal
  - Evreux - CH, Évreux
  - Flers - CH, Flers
  - CHICAS Site de Gap, Gap
  - CHRU Grenoble, Grenoble
  - Saint Omer - CHI, Helfaut
  - Jonzac - CH, Jonzac
  - La Roche Sur Yon - CH, La Roche-sur-Yon
  - Le Havre - HPE, Le Havre
  - Le Mans - Centre Hospitalier, Le Mans
  - Le Mans - Clinique Victor Hugo, Le Mans
  - CH Dr Schaffner de Lens, Lens
  - Liévin - polyclinique de Riaumont, Liévin
  - CHU (Hôpital Calmette) - Pneumologie, Lille
  - Lille - Hôpital Calmette, Lille
  - Limoges - Hôpital du Cluzeau, Limoges
  - CH de Longjumeau, Longjumeau
  - Lorient - CHBS, Lorient
  - Clinique des 4 Pavillons, Lormont
  - Lyon - Clinique Mutualiste, Lyon
  - Clinique Mutualiste Eugène André, Lyon
  - HIA Desgenettes, Lyon
  - Hôpital de la Croix Rousse, Lyon
  - Lyon - Hôpital Louis Pradel (Pneumologie), Lyon
  - Mantes La Jolie - CH, Mantes-la-Jolie
  - Marseille - Hôpital Sainte Marguerite, Marseille
  - Marseille - CRLCC, Marseille
  - Polyclinique du Parc, Maubeuge
  - Meaux - CH, Meaux
  - Metz - CHR, Metz
  - Metz - Clinique Claude Bernard, Metz
  - Metz - Belle Isle, Metz
  - Mont de Marsan - CH, Mont-de-Marsan
  - Montpellier - Clinique Clémentville, Montpellier
  - Montpellier - CHRU, Montpellier
  - Moulins - CH, Moulins
  - Mulhouse - CH, Mulhouse
  - CHU Nancy, Nancy
  - Nancy - Polyclinique Gentilly, Nancy
  - Nanterre - CH, Nanterre
  - Nantes - Centre René Gauducheau, Nantes
  - Hôpital Laënnec - CHU de Nantes, Nantes
  - Narbonne - Polyclinique Le Languedoc, Narbonne
  - Neuilly - Hôpital Américain de Paris, Neuilly
  - Nevers - CH, Nevers
  - Nice - CAC, Nice
  - Nîmes - Clinique Valdegour, Nîmes
  - CHU, Nîmes
  - Orléans - CH, Orléans
  - Paris - Saint Louis, Paris
  - Paris - hôpital Saint-Antoine, Paris
  - GH Paris Saint-Joseph, Paris
  - Hôpital Bichat - Claude - Bernard, Paris
  - Hôpital du Val de Grâce, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Tenon, Paris
  - Paris - Curie, Paris
  - Pau - CH, Pau
  - Perpignan - Centre Catalan d'Oncologie, Perpignan
  - Perpignan - Ch, Perpignan
  - CH de Périgueux, Périgueux
  - Lyon Sud, Pierre-Bénite
  - CHU, Poitiers
  - Pontoise - CH, Pontoise
  - Reims - CHU, Reims
  - Reims - CRLCC, Reims
  - Rennes - CHU, Rennes
  - CHG de Roanne, Roanne
  - Rodez - CH, Rodez
  - Roncq - Clinique Saint-Roch, Roncq
  - Roubaix - CH, Roubaix
  - Rouen - CHU, Rouen
  - Centre Frederic Joliot, Rouen
  - Saint Brieuc - CHG, Saint-Brieuc
  - Saint Nazaire - Centre Etienne Dolet, Saint-Nazaire
  - Saint-Nazaire - CH, Saint-Nazaire
  - Saint Priest en Jarez - ICL, Saint-Priest-en-Jarez
  - Saint Quentin - CH, Saint-Quentin
  - Saverne - CH, Saverne
  - Senlis - CH, Senlis
  - Saint-Malo - CH, St-Malo
  - Strasbourg - NHC, Strasbourg
  - Suresnes - Hopital Foch, Suresnes
  - Thonon les bains, Thonon-les-Bains
  - Toulon - CHI, Toulon
  - Toulon - HIA, Toulon
  - Clinique Saint Jean du Languedoc, Toulouse
  - Toulouse - CHU Larrey, Toulouse
  - Toulouse - Clinique Pasteur, Toulouse
  - Tours - CHU, Tours
  - Troyes - CH, Troyes
  - Valenciennes - Clinique, Valenciennes
  - Verdun - CHG, Verdun
  - Vesoul - CHI, Vesoul
  - CHI de la Haute-Saône - Pneumologie, Vesoul
  - Clinique Mutualiste Les Portes du Sud, Vénissieux
  - Vienne - CH, Vienne
  - Villejuif - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blons H, Oudart JB, Merlio JP, Debieuvre D, de Fraipont F, Audigier-Valette C, Escande F, Hominal S, Bringuier PP, Fraboulet-Moreau S, Ouafik L, Moro-Sibilot D, Lemoine A, Langlais A, Missy P, Morin F, Souquet PJ, Barlesi F, Cadranel J, Beau-Faller M; French Cooperative Thoracic Intergroup (IFCT). PTEN, ATM, IDH1 mutations and MAPK pathway activation as modulators of PFS and OS in patients treated by first line EGFR TKI, an ancillary study of the French Cooperative Thoracic Intergroup (IFCT) Biomarkers France project. Lung Cancer. 2021 Jan;151:69-75. doi: 10.1016/j.lungcan.2020.11.008. Epub 2020 Nov 13. PMID 33248711
- [Background] Beau-Faller M, Pencreach E, Leduc C, Blons H, Merlio JP, Bringuier PP, de Fraipont F, Escande F, Lemoine A, Ouafik L, Denis M, Hofman P, Lacave R, Melaabi S, Langlais A, Missy P, Morin F, Moro-Sibilot D, Barlesi F, Cadranel J; French Cooperative Thoracic Intergroup (IFCT). Independent prognostic value of ultra-sensitive quantification of tumor pre-treatment T790M subclones in EGFR mutated non-small cell lung cancer (NSCLC) treated by first/second generation TKI, depends on variant allele frequency (VAF): Results of the French cooperative thoracic intergroup (IFCT) biomarkers France project. Lung Cancer. 2020 Feb;140:19-26. doi: 10.1016/j.lungcan.2019.10.013. Epub 2019 Nov 15. PMID 31841714
- [Background] Leduc C, Merlio JP, Besse B, Blons H, Debieuvre D, Bringuier PP, Monnet I, Rouquette I, Fraboulet-Moreau S, Lemoine A, Pouessel D, Mosser J, Vaylet F, Langlais A, Missy P, Morin F, Moro-Sibilot D, Cadranel J, Barlesi F, Beau-Faller M; French Cooperative Thoracic Intergroup (IFCT). Clinical and molecular characteristics of non-small-cell lung cancer (NSCLC) harboring EGFR mutation: results of the nationwide French Cooperative Thoracic Intergroup (IFCT) program. Ann Oncol. 2017 Nov 1;28(11):2715-2724. doi: 10.1093/annonc/mdx404. PMID 28945865
- [Background] Kembou Nzale S, Weeks WB, Ouafik L, Rouquette I, Beau-Faller M, Lemoine A, Bringuier PP, Le Coroller Soriano AG, Barlesi F, Ventelou B. Inequity in access to personalized medicine in France: Evidences from analysis of geo variations in the access to molecular profiling among advanced non-small-cell lung cancer patients: Results from the IFCT Biomarkers France Study. PLoS One. 2020 Jul 1;15(7):e0234387. doi: 10.1371/journal.pone.0234387. eCollection 2020. PMID 32609781
- [Background] Mordant P MD, PhD, Brosseau S, Milleron B, Santelmo N, Fraboulet-Moreau S, Besse B, Langlais A, Gossot D, Thomas PA, Pujol JL, Ricordel C, Madelaine J, Lamy R, Audigier-Valette C, Missy P, Blons H, Barlesi F, Westeel V; French Cooperative Thoracic Intergroup (IFCT). Outcome of Patients With Resected Early-Stage Non-small Cell Lung Cancer and EGFR Mutations: Results From the IFCT Biomarkers France Study. Clin Lung Cancer. 2023 Jan;24(1):1-10. doi: 10.1016/j.cllc.2022.08.013. Epub 2022 Aug 29. PMID 36180314
- [Background] Guibert N, Barlesi F, Descourt R, Lena H, Besse B, Beau-Faller M, Mosser J, Pichon E, Merlio JP, Ouafik L, Guichard F, Mastroianni B, Moreau L, Wdowik A, Sabourin JC, Lemoine A, Missy P, Langlais A, Moro-Sibilot D, Mazieres J. Characteristics and Outcomes of Patients with Lung Cancer Harboring Multiple Molecular Alterations: Results from the IFCT Study Biomarkers France. J Thorac Oncol. 2017 Jun;12(6):963-973. doi: 10.1016/j.jtho.2017.02.001. Epub 2017 Feb 9. PMID 28189832
- [Background] Couraud S, Barlesi F, Fontaine-Deraluelle C, Debieuvre D, Merlio JP, Moreau L, Beau-Faller M, Veillon R, Mosser J, Al Freijat F, Bringuier PP, Lena H, Ouafik L, Westeel V, Morel A, Audigier-Valette C, Missy P, Langlais A, Morin F, Souquet PJ, Planchard D; Biomarkers France Contributors. Clinical outcomes of non-small-cell lung cancer patients with BRAF mutations: results from the French Cooperative Thoracic Intergroup biomarkers France study. Eur J Cancer. 2019 Jul;116:86-97. doi: 10.1016/j.ejca.2019.04.016. Epub 2019 Jun 8. PMID 31181537
- [Background] Ruppert AM, Beau-Faller M, Debieuvre D, Ouafik L, Westeel V, Rouquette I, Mazieres J, Bringuier PP, Monnet I, Escande F, Ricordel C, Merlio JP, Janicot H, Lemoine A, Foucher P, Poudenx M, Morin F, Langlais A, Souquet PJ, Barlesi F, Wislez M. Outcomes of Patients With Advanced NSCLC From the Intergroupe Francophone de Cancerologie Thoracique Biomarkers France Study by KRAS Mutation Subtypes. JTO Clin Res Rep. 2020 May 15;1(3):100052. doi: 10.1016/j.jtocrr.2020.100052. eCollection 2020 Sep. PMID 34589947
- [Background] Tomasini P, Brosseau S, Mazieres J, Merlio JP, Beau-Faller M, Mosser J, Wislez M, Ouafik L, Besse B, Rouquette I, Debieuvre D, Escande F, Westeel V, Audigier-Valette C, Missy P, Langlais A, Morin F, Moro-Sibilot D, Zalcman G, Barlesi F. EGFR tyrosine kinase inhibitors versus chemotherapy in EGFR wild-type pre-treated advanced nonsmall cell lung cancer in daily practice. Eur Respir J. 2017 Aug 10;50(2):1700514. doi: 10.1183/13993003.00514-2017. Print 2017 Aug. PMID 28798090
- [Result] Barlesi F, Mazieres J, Merlio JP, Debieuvre D, Mosser J, Lena H, Ouafik L, Besse B, Rouquette I, Westeel V, Escande F, Monnet I, Lemoine A, Veillon R, Blons H, Audigier-Valette C, Bringuier PP, Lamy R, Beau-Faller M, Pujol JL, Sabourin JC, Penault-Llorca F, Denis MG, Lantuejoul S, Morin F, Tran Q, Missy P, Langlais A, Milleron B, Cadranel J, Soria JC, Zalcman G; Biomarkers France contributors. Routine molecular profiling of patients with advanced non-small-cell lung cancer: results of a 1-year nationwide programme of the French Cooperative Thoracic Intergroup (IFCT). Lancet. 2016 Apr 2;387(10026):1415-1426. doi: 10.1016/S0140-6736(16)00004-0. Epub 2016 Jan 15. PMID 26777916
- See also: IFCT official website — http://www.ifct.fr/